CLINICAL TRIAL: NCT02382926
Title: Capacitive Electrocardiography in the Driver's Seat and Elevation of Vital Signs Via Camera During Cardiac Rehabilitation
Brief Title: Reha Drive: Capacitive Electrocardiography in Car Seat in Cardiological Patients
Acronym: RehaDrivecECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: RWTH Aachen Institute of Medical Information Technology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CTC-A 14-053
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Cardiac Events
Keywords: capacitive electrocardiography; Eulerian Magnification Method
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- contactless heart-, breathing rate, ECG (Experimental)
  Interventions: Other: Capacitive ECG and contactless heart and breathing rate measurements via camera

INTERVENTIONS:
Other: Capacitive ECG and contactless heart and breathing rate measurements via camera — During a 30 minute driving simulation cardiologic patients in rehabilitation undergo capacitive ECG measurements via sensors in the car seat as well as heart and breathing rate measurements via camera according to the Eulerian Magnification Method.

SUMMARY:
In this trial contactless heart rate, electrocardiography and breathing rate measurements are elevated during car simulation in cardiac rehabilitation via automotive sensors and camera.

DETAILED DESCRIPTION:
Increasing number of elderly people with cardiovascular diseases and the wish to drive a car need recommendations corresponding to their fitness of driving during cardiac rehabilitation. Little trial data are known, only a position paper of the German Cardiac Society (DGK) of 2010 discusses the aptitude of driving a car of cardiovascular patients on experience. For judgement and recommendations automotive monitoring via contactless sensors might be helpful. Therefore while "driving" in a simulator distinct heart circulation situations will be created. Vital signs will be measured via long term electrocardiography (ECG) in comparison to contactless capacitive ECG (cECG) measurements via embedded sensors in the car seat as well as heart rate and breathing rate measurements via camera.

ELIGIBILITY:
Inclusion Criteria:

* cardiologic diseases after acute event (e. g. myocard infarction, bypass surgery)
* rehabilitation in clinic "An der Rosenquelle"

Exclusion Criteria:

* dementia
* lack of language ability
* pregnancy
* implanted electric devices (as e.g. heart pacemaker, inverted cardiodefibrillator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
arrhythmia | 30 minutes
  feasibility of cECG data for example as arrhythmia, tachycardia in comparison to long term ECG data

SECONDARY OUTCOMES:
Heart rate via contactless camera | 30 minutes
  feasibility of heart rate measurements according to the Eulerian Magnification Method in comparison to standard measurement data

OTHER OUTCOMES:
Breathing rate via contactless camera | 30 minutes
  feasibility of breathing rate measurements according to the Eulerian Magnification Method in comparison to standard measurement data

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Reith, MD, Principal Investigator — University Hospital Aachen, Clinic of Cardiology, Angiology, Pneumology and Intensive Care Medicine
Locations (2):
- Germany (2):
  - Clinic of Rehabilitation "An der Rosenquelle", Kurbrunnenstreet 5, Aachen, North Rhine-Westphalia
  - University Hospital Aachen, Department of Cardiology, Angiology, Pneumology and Intensive Medicine, Aachen, North Rhine-Westphalia